CLINICAL TRIAL: NCT01138306
Title: Implications of s-SHIP Expression and SHIP Alterations in AML
Brief Title: Biomarkers in Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B5; COG-AAML10B5 (Other: Children's Oncology Group); CDR0000671462 (Other: Clinical Trials.gov); NCI-2011-02223 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Gene Expression Profiling; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the extent and prognostic implications of variable s-SHIP expression and SHIP gene mutations in pediatric patients with acute myeloid leukemia.
* Determine the effects of aberrant s-SHIP expression on the PI3K/Akt pathway in these patients via electrochemiluminescence and phosphospecific flow cytometry assays.

OUTLINE: RNA samples are analyzed for variable s-SHIP expression and are screened for SHIP mutations. Cryopreserved cells (with known high- or low-s-SHIP expression) are analyzed for the levels of various components of the PI3K/Akt pathway via electrochemiluminescence and phosphospecific flow cytometry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 149 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
Overall survival
Relapse rate

CONTACTS AND LOCATIONS:
Overall Officials: Phoenix Ho, MD, Principal Investigator — Fred Hutchinson Cancer Center